CLINICAL TRIAL: NCT06422429
Title: Study on the Regulatory Effects of Personalized Innovative Youtiao Intervention on Nutritional Health
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yu Zhang (Other)
Responsible Party: Sponsor-Investigator, Yu Zhang, professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT_PI Youtiao
Record Dates: First submitted 2024-01-17; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-01

CONDITIONS: Metabolism and Nutrition Disorder
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): traditional Youtiao
  Interventions: Drug: Traditional deep-fried Youtiao
- Intervention group (Experimental): Personalised and innovative Youtiao
  Interventions: Drug: PI Youtiao

INTERVENTIONS:
Drug: Traditional deep-fried Youtiao — 45g 4 times a week for 4 months
  Arms: Control group
Drug: PI Youtiao — 45g 4 times a week for 4 months
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to investigate the effects of personalized innovative fritters on the nutritional health of overweight and obese individuals aged 40 to 70 years. The main questions it aims to answer are:

* How does consuming personalized innovative fritters affect the nutritional health of overweight and obese individuals?
* What is the mechanism underlying the impact of personalized innovative oil bars on nutritional health?

Participants will be randomly assigned to one of two groups: a trial group consuming personalized innovative fritters and a control group consuming traditional fritters with equal energy content. Over the course of 6 months, participants will undergo two phases of intervention separated by a two-month washout period. During the intervention, participants will be assessed comprehensively for sensory ratings and nutritional health status through biological indicators, physical examinations, and other relevant measures.

Researchers will compare the trial group to the control group to determine if personalized innovative fritters lead to improvements in nutritional health compared to traditional fritters.

DETAILED DESCRIPTION:
Participants entered the trial with a 1-week equilibration period during which baked and fried foods were prohibited. The test group will consume personalised innovative Youtiao and the control group will uniformly consume traditional Youtiao of equal energy, 45 g 4 times per week for 8 weeks, during which time we will periodically measure biological indicators and collect biological samples to gain insight into the effects of the personalised innovative Youtiao on the participants. After completion of the 8-week intervention, a washout phase is entered. During this phase, participants will no longer ingest the Youtiao to see how they trend after stopping the intervention. Participants then enter the second phase of the trial, where the intervention process described above is continued with appropriate consumption adjustments based on the initial results of the first phase of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-70 years old (women need to be menopausal);
* BMI>24 kg/m2;
* Consumption of fritters more than once a week.

Exclusion Criteria:

* history of diabetes mellitus, cardiovascular disease, dyslipidaemia, renal disease, -
* liver disease or cancer;
* surgical treatment within 3 months;
* allergy/intolerance to the study food or any of its ingredients;
* breastfeeding or pregnancy;
* >10% weight loss in the past 6 months;
* smoking or alcohol abuse;
* participation in another clinical study within the past 6 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  The investigators will measure HbA1c in blood samples before and after treatment.
Change in blood glucose from baseline | 6 months
  The investigators will measure fasting plasma glucose levels in blood samples before and after treatment.

SECONDARY OUTCOMES:
Change in blood lipids from baseline | 6 months
  The investigators will measure Triglycerides (TG), total cholesterol (TC), LDL-C, and HDL-C levels in blood samples before and after treatment.